CLINICAL TRIAL: NCT07071714
Title: An Open, Multicenter Phase II Study of SHR-8068 Injection in Combination With Anti-tumor Therapies in Colorectal Cancer
Brief Title: A Phase II Study of SHR-8068 Injection in Combination With Anti-tumor Therapies in Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-8068-206
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A Group (Experimental)
  Interventions: Drug: SHR-8068 Injection; Drug: Adebrelimab Injection
- Part B Group (Experimental)
  Interventions: Drug: SHR-8068 Injection; Drug: Adebrelimab Injection; Drug: Bevacizumab Injection

INTERVENTIONS:
Drug: SHR-8068 Injection — SHR-8068 injection.
Drug: Adebrelimab Injection — Adebrelimab injection.
Drug: Bevacizumab Injection — Bevacizumab injection.
  Arms: Part B Group

SUMMARY:
The study is being conducted to evaluate the safety, tolerability and efficacy of SHR-8068 injection in combination with anti-tumor therapies in subjects with colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily agree to participate in the trial and sign a written informed consent form.
2. Male or female ≥ 18 years old and ≤75 years old.
3. ECOG performance status of 0-1.
4. Part A with a life expectancy of ≥2 years. Part B with a life expectancy of ≥12 weeks.
5. Need to provided tumor tissue samples for genetic testing.

Exclusion Criteria:

1. Part B: Accompanied by untreated or active central nervous system (CNS) metastases. Subjects with a history or current history of meningeal metastasis.
2. Part B: Systemic antitumor therapy was received 4 weeks before the start of the study.
3. Part B: Palliative radiotherapy was completed within 14 days before the first dose.
4. Toxicity and/or complications from previous interventions did not return to NCI-CTCAE level ≤1 or exclusion criteria.
5. Subjects with known or suspected interstitial pneumonia.
6. Moderate or severe ascites with clinical symptoms; Uncontrolled or moderate or higher pleural effusion or pericardial effusion.
7. Have poorly controlled or severe cardiovascular disease.
8. Subjects with active hepatitis B or active hepatitis C.
9. A history of immunodeficiency, including a positive HIV test, other acquired or congenital immunodeficiency disorders, or a history of organ transplantation.
10. The presence of uncontrolled mental illness and other conditions known to affect the completion of the study process, such as alcohol, drug or substance abuse, and criminal detention.
11. Any other factors that may increase the risk of participating in the study, interfere with the study results, or make participation in the study inappropriate as judged by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2031-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | About 7 months.
Progression Free Survival (PFS) | About 18 months.

SECONDARY OUTCOMES:
Clinical Complete Response (cCR) | About 60 months.
Disease Free Survival (DFS) | About 60 months.
Event Free Survival (EFS） | About 60 months.
Overall Survival (OS) | About 60 months.
Duration of Response (DoR) | About 18 months.
Overall Response Rate (ORR) | About 18 months.
Disease Control Rate (DCR) | About 18 months.
Adverse Events (AEs) | Up to about 18 months.

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided